CLINICAL TRIAL: NCT00946543
Title: A Phase I Dose Escalation Study of the Use of Intensity Modulated Radiotherapy (IMRT) to Treat Prostate and Pelvic Nodes in Patients With Prostate Cancer - Pelvic IMRT for Prostate Cancer
Brief Title: Intensity-Modulated Radiation Therapy in Treating Patients With Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000601695; RMNHS-1766; EU-20869
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-07

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Radiation: hypofractionated radiation therapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the best dose of intensity-modulated radiation therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the feasibility of delivering hypofractionated intensity-modulated radiotherapy to the prostate and pelvic nodes of patients with prostate cancer.
* To determine the optimal dose level of this treatment regimen to be used in future studies.

OUTLINE: Patients are stratified according to small bowel total volume (low small bowel volume < 450 cc vs high small bowel volume ≥ 450 cc).

Patients undergo hypofractionated intensity-modulated radiotherapy to the prostate and pelvis for 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 5 years and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer meeting 1 of the following criteria:

  * Stage T3b/T4 disease or radiological or pathological pelvic nodal metastases
  * Localized disease (stage pT2-T4) with > 30% estimated risk of pelvic nodal metastases
  * High-risk (Gleason score ≥ 8 or ≥ 2 risk factors) or very high-risk disease according to the National Collaborative Cancer Network (NCCN)
  * Has undergone prostatectomy AND has stage T2-T3a, N0 disease with extensive high-risk disease (Gleason score ≥ 8) or seminal vesicle or lymph node involvement
* Candidate for radical radiotherapy

PATIENT CHARACTERISTICS:

* No inflammatory bowel disease or other small bowel disease

PRIOR CONCURRENT THERAPY:

* No prior pelvic radiotherapy or surgery (excluding prostatectomy)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2000-03; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Late RTOG radiotherapy toxicity as assessed at 6, 12, 18, and 24 months and then annually thereafter

SECONDARY OUTCOMES:
Overall survival
Local control
PSA control
Acute side effects as assessed weekly by the RTOG scoring system
Quality of life
Patterns of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: David P. Dearnaley, MD, FRCP, FRCR, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Institute of Cancer Research - Chelsea, London, England
  - Institute of Cancer Research - Sutton, Sutton, England
  - Royal Marsden - Surrey, Sutton, England

REFERENCES:
- [Derived] Fernandez-Mateos J, Cresswell GD, Trahearn N, Webb K, Sakr C, Lampis A, Stuttle C, Corbishley CM, Stavrinides V, Zapata L, Spiteri I, Heide T, Gallagher L, James C, Ramazzotti D, Gao A, Kote-Jarai Z, Acar A, Truelove L, Proszek P, Murray J, Reid A, Wilkins A, Hubank M, Eeles R, Dearnaley D, Sottoriva A. Tumor evolution metrics predict recurrence beyond 10 years in locally advanced prostate cancer. Nat Cancer. 2024 Sep;5(9):1334-1351. doi: 10.1038/s43018-024-00787-0. Epub 2024 Jul 12. PMID 38997466